CLINICAL TRIAL: NCT00801424
Title: Randomized Clinical Study for Core and Topical Warming of the Open Wound Cavity With Warmed Humidified CO2 Versus Control in Colon Surgery
Brief Title: Warmed Humidified Carbon Dioxide (CO2) for Open Surgery
Acronym: S2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Jan van der Linden, Professor, Karolinska Institute / Karolinska University Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2008/1258-31-4
Record Dates: First submitted 2008-12-01; First posted 2008-12-03 (Estimated); Last update posted 2010-10-04 (Estimated); Status verified 2010-10

CONDITIONS: Hypothermia
Keywords: abdominal surgery; hypothermia; wound dessication; warming
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- standard heating (Experimental): Standard intraoperative warming measures including heated sheets, heating with forced warmed air, warming of fluids, and insulation of limbs and head.
  Interventions: Device: humidified warmed CO2

INTERVENTIONS:
Device: humidified warmed CO2 — Additional insufflation of humidified carbon dioxide (approx. 36-37ºC, approx. 80-100% relative humidity) via a humidifier with a heated tube (Fisher&Paykel) connected to a gas diffuser (Cardia Innovation AB) that is able to create a local atmosphere of 100% carbon dioxide (humidified) in the wound cavity

SUMMARY:
Eighty adult patients undergoing open colon surgery will be randomized to either:

1. standard warming measures including heating sheets, warming of fluids, and insulation of limbs and head, or to
2. additional insufflation of humidified carbon dioxide (approx. 36-37ºC, approx. 80-100% relative humidity) via a humidifier with a heated tube (Fisher&Paykel) connected to a gas diffuser (Cardia Innovation AB) that is able to create a local atmosphere of 100% carbon dioxide (humidified ) in the open wound cavity.

PRIMARY AIM The primary aim of this study is to evaluate if humidified carbon dioxide insufflated into an open surgical wound can be used to warm the core, the open wound cavity, and the wound edges during major abdominal surgery.

SECONDARY AIMS Secondary aims are to evaluate possible differences between the groups regarding complications and clinical differences including histological signs of desiccation injury of peritoneal samples, time to extubation, core temperature after surgery, ICU stay, bleeding volume, hospital stay, postoperative pain, infections, shivering, postoperative signs of restored bowel function including bowel movements, flatus, and first meal.

DETAILED DESCRIPTION:
Eighty patients undergoing open colon surgery will be randomized to either standard warming measures including heating sheets, warming of fluids, and insulation of limbs and head or to additional insufflation of humidified carbon dioxide (approx. 36-37ºC, approx. 80-100% relative humidity) via a humidifier with a heated tube (Fisher&Paykel) connected to a gas diffuser (Cardia Innovation AB) that is able to create a local atmosphere of 100% carbon dioxide (humidified) in the wound cavity.

Wound temperatures will be measured every 10 minutes with an infra-red camera positioned approximately 1m above the wound with a camera support. Wound areas and wound edges of stored images will be delineated with a soft ware program. Peritoneal samples (3x3x1mm) will be taken at start of the operation, after 30 minutes and before closure of the abdomen. The samples will immediately be stored in RNA-later solution, and deep frozen for later analysis of epithelial (peritoneal) and endothelial function/tissue damage.

ELIGIBILITY:
Inclusion Criteria:

* major open abdominal surgery (colon surgery) in adults
* patient signed informed consent

Exclusion Criteria:

* acute surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Temperature of the core, the open wound cavity including the wound edges during major abdominal surgery | duration surgery up to 12 hours

SECONDARY OUTCOMES:
Time to extubation | up to 30 days after surgery
Histological signs of dessication injury of peritoneal samples | duration surgery up to 12 hours
ICU stay | up to 30 days after surgery
Pain and need of analgesia | up to 30 days after surgery
Restoration of bowel function after surgery including flatus, bowel movements, and first meal | up to 30 days after surgery
Postoperative infections including pneumonia and surgical site infection | up to 30 days after surgery
Postoperative shivering | up to 24 hours after surgery
Suture removal | up to 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jan A van der Linden, MD PhD, Principal Investigator — Karolinska Institute / Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Background] Persson M, van der Linden J. Intraoperative CO2 insufflation can decrease the risk of surgical site infection. Med Hypotheses. 2008;71(1):8-13. doi: 10.1016/j.mehy.2007.12.016. Epub 2008 Mar 4. PMID 18304752
- [Background] Persson M, van der Linden J. Can wound desiccation be averted during cardiac surgery? An experimental study. Anesth Analg. 2005 Feb;100(2):315-320. doi: 10.1213/01.ANE.0000140243.97570.DE. PMID 15673849
- [Background] Persson M, Elmqvist H, van der Linden J. Topical humidified carbon dioxide to keep the open surgical wound warm: the greenhouse effect revisited. Anesthesiology. 2004 Oct;101(4):945-9. doi: 10.1097/00000542-200410000-00020. PMID 15448528
- [Background] Persson M, Svenarud P, Flock JI, van der Linden J. Carbon dioxide inhibits the growth rate of Staphylococcus aureus at body temperature. Surg Endosc. 2005 Jan;19(1):91-4. doi: 10.1007/s00464-003-9334-z. Epub 2004 Nov 11. PMID 15529188
- [Background] Persson M, van der Linden J. Wound ventilation with ultraclean air for prevention of direct airborne contamination during surgery. Infect Control Hosp Epidemiol. 2004 Apr;25(4):297-301. doi: 10.1086/502395. PMID 15108726
- [Background] Persson M, van der Linden J. Wound ventilation with carbon dioxide: a simple method to prevent direct airborne contamination during cardiac surgery? J Hosp Infect. 2004 Feb;56(2):131-6. doi: 10.1016/j.jhin.2003.10.013. PMID 15019225
- [Background] Persson M, Van Der Linden J. De-airing of a cardiothoracic wound cavity model with carbon dioxide: theory and comparison of a gas diffuser with conventional tubes. J Cardiothorac Vasc Anesth. 2003 Jun;17(3):329-35. doi: 10.1016/s1053-0770(03)00050-8. PMID 12827581
- [Background] Svenarud P, Persson M, Van Der Linden J. Efficiency of a gas diffuser and influence of suction in carbon dioxide deairing of a cardiothoracic wound cavity model. J Thorac Cardiovasc Surg. 2003 May;125(5):1043-9. doi: 10.1067/mtc.2003.50. PMID 12771877
- [Background] Svenarud P, Persson M, van der Linden J. Intermittent or continuous carbon dioxide insufflation for de-airing of the cardiothoracic wound cavity? An experimental study with a new gas-diffuser. Anesth Analg. 2003 Feb;96(2):321-7, table of contents. doi: 10.1097/00000539-200302000-00005. PMID 12538172
- [Background] Hannenberg AA, Sessler DI. Improving perioperative temperature management. Anesth Analg. 2008 Nov;107(5):1454-7. doi: 10.1213/ane.0b013e318181f6f2. No abstract available. PMID 18931198
- [Background] Sessler DI. Temperature monitoring and perioperative thermoregulation. Anesthesiology. 2008 Aug;109(2):318-38. doi: 10.1097/ALN.0b013e31817f6d76. PMID 18648241
- [Background] Insler SR, Sessler DI. Perioperative thermoregulation and temperature monitoring. Anesthesiol Clin. 2006 Dec;24(4):823-37. doi: 10.1016/j.atc.2006.09.001. PMID 17342966
- [Background] Sessler DI. Non-pharmacologic prevention of surgical wound infection. Anesthesiol Clin. 2006 Jun;24(2):279-97. doi: 10.1016/j.atc.2006.01.005. PMID 16927930